CLINICAL TRIAL: NCT05659134
Title: Comparison of Alfredson Eccentric and Silbernagel Concentric-eccentric Therapeutical Protocol in Competitive Athletes With Chronic Achilles Tendinopathy
Brief Title: Comparison of Alfredson and Silbernagel Protocol in Competitive Athletes With Achilles Tendinopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kryštof Voleský, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 254/21
Record Dates: First submitted 2022-11-14; First posted 2022-12-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Achilles Tendinopathy; Tendon Injuries; Tendon Thickening; Pain, Chronic
Keywords: Achilles tendinopathy; VISA-A; Ultrasound; Stiffness; Competitive athletes; Exercise therapy; Alfredson protocol; Silbernagel protocol
MeSH Terms: conditions — Tendon Injuries; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alfredson group (A) (Active Comparator): Participants allocated to the Alfredson exercise program were instructed to exercise twice a day on both legs for 12 months. They performed concentric calf rises (CR) on both legs up and eccentric CR on one leg down.
  The protocol contained 15 repetitions and 3 sets on each leg with extended and flexed knee. One session contained 45 reps in the flexed position and 45 reps in the extended position, the total daily number of reps was 180. At the start, the exercises were performed with body weight. Participants could progress by adding the 5, 10 and 15 kg, if they met the criteria. The criteria for adding weight was at least one week of training at the same weight and no disabling pain during or after the exercise during the week.
  Interventions: Other: Alfredson protocol
- Silbernagel group (B) (Active Comparator): Participants allocated to the Silbernagel exercise program were instructed to exercise every day with exception of the first week (every other day) for 12 months. The protocol contained 4 phases, which were based on a variety of CR exercises.
  The protocol contained concentric and eccentric CR on both legs, CR on one leg, CR in sitting, CR on the step, CR without step, quick rebound CR, CR with added weight and hops on the forefoot.
  The daily number of reps for 1st phase was 135, for the 2nd phase was 240, for the 3rd phase was 255 and for the 4th phase was 150. It's performed with body weight, added weight and plyometric loading progressively through all phases (maximal added weight is 15 kilos). To progress to the next phase participant needs to reach pain intensity during and after exercise under 5 from the 10 on the visual analogue scale, morning stiffness should not increase as well as pain during the week.
  Interventions: Other: Silbernagel protocol

INTERVENTIONS:
Other: Alfredson protocol — Alfredson eccentric therapeutical protocol.
  Arms: Alfredson group (A)
Other: Silbernagel protocol — Silbernagel concentric-eccentric protocol.
  Arms: Silbernagel group (B)

SUMMARY:
A 6-week randomized clinical trial (RCT) with a 46-week follow-up compared the effect of Alfredson and Silbernagel eccentric programs for the treatment of AT. The primary outcome was a change in the Victorian Institute of Sport Assessment - Achilles (VISA-A) scale from baseline to 12 months. The study was approved by the Ethics Committee of the Faculty of Physical Education and Sport, Charles University (Project number: 254/2021). All participants provided written informed consent before participation.

ELIGIBILITY:
Inclusion criteria:

* Athletes performing track and field, tennis or football at the competitive level
* Age 18 to 40 years
* Unilateral Achilles tendinopathy
* Pain lasting more than 2 months
* Diagnosis of Achilles tendinopathy established by pain on function at the Achilles region and ultrasound assessment (tendon thickening, swollen tendon) by one researcher
* Participants trained at least 3 times per week before the onset of Achilles tendinopathy
* Less than 3 months without training and less than 6 months from the last competition/match
* Wish to return to original sport level
* Willing to stop with other treatments 2 weeks before the start of the clinical trial

Exclusion criteria:

* Achilles tendon rupture in past
* Corticosteroid injection in Achilles tendon region in last 6 months
* Having other lower limb musculoskeletal injuries or surgery in the last 6 months (e.g., muscle rupture, bone fracture)
* Having a neurological, systemic or autoimmune disease (e.g., neuropathy, type 1 diabetes, rheumatoid arthritis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles (VISA-A) | 1 year
  The VISA-A questionnaire is the most commonly used outcome in clinical trials of Achilles tendinopathy treatment with proven reliability and validity. It consists of eight questions covering pain, function, daily living and sports activities. The score ranges from 0-100 where 0 means disability (impairment of function and pain of Achilles tendon) and 100 represents no disability.

SECONDARY OUTCOMES:
Biomechanical properties - stiffness | 6 weeks
  Achilles tendon stiffness (N/m) is a measure of the biomechanical response of the Achilles tendon tissue. Stiffness was assessed by MyotonPro (Myoton AS), which has been shown as a valid and reliable measurement tool of Achilles tendon mechanical properties in the clinical setting.
Structure - micromorphology | 6 weeks
  Fibre organisation analysis of PSFR (mmˆ-1).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Education and Sport at Charles University, Prague, Prague 6, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scott A, Squier K, Alfredson H, Bahr R, Cook JL, Coombes B, de Vos RJ, Fu SN, Grimaldi A, Lewis JS, Maffulli N, Magnusson SP, Malliaras P, Mc Auliffe S, Oei EHG, Purdam CR, Rees JD, Rio EK, Gravare Silbernagel K, Speed C, Weir A, Wolf JM, Akker-Scheek IVD, Vicenzino BT, Zwerver J. ICON 2019: International Scientific Tendinopathy Symposium Consensus: Clinical Terminology. Br J Sports Med. 2020 Mar;54(5):260-262. doi: 10.1136/bjsports-2019-100885. Epub 2019 Aug 9. No abstract available. PMID 31399426
- [Background] Wang Y, Zhou H, Nie Z, Cui S. Prevalence of Achilles tendinopathy in physical exercise: A systematic review and meta-analysis. Sports Med Health Sci. 2022 Mar 28;4(3):152-159. doi: 10.1016/j.smhs.2022.03.003. eCollection 2022 Sep. PMID 36090915
- [Background] Sleeswijk Visser TSO, van der Vlist AC, van Oosterom RF, van Veldhoven P, Verhaar JAN, de Vos RJ. Impact of chronic Achilles tendinopathy on health-related quality of life, work performance, healthcare utilisation and costs. BMJ Open Sport Exerc Med. 2021 Mar 26;7(1):e001023. doi: 10.1136/bmjsem-2020-001023. eCollection 2021. PMID 33868707
- [Background] van der Plas A, de Jonge S, de Vos RJ, van der Heide HJ, Verhaar JA, Weir A, Tol JL. A 5-year follow-up study of Alfredson's heel-drop exercise programme in chronic midportion Achilles tendinopathy. Br J Sports Med. 2012 Mar;46(3):214-8. doi: 10.1136/bjsports-2011-090035. Epub 2011 Nov 10. PMID 22075719
- [Background] van der Vlist AC, Winters M, Weir A, Ardern CL, Welton NJ, Caldwell DM, Verhaar JAN, de Vos RJ. Which treatment is most effective for patients with Achilles tendinopathy? A living systematic review with network meta-analysis of 29 randomised controlled trials. Br J Sports Med. 2021 Mar;55(5):249-256. doi: 10.1136/bjsports-2019-101872. Epub 2020 Jun 10. PMID 32522732
- [Background] Silbernagel KG, Crossley KM. A Proposed Return-to-Sport Program for Patients With Midportion Achilles Tendinopathy: Rationale and Implementation. J Orthop Sports Phys Ther. 2015 Nov;45(11):876-86. doi: 10.2519/jospt.2015.5885. Epub 2015 Sep 21. PMID 26390272
- [Background] Breda SJ, Oei EHG, Zwerver J, Visser E, Waarsing E, Krestin GP, de Vos RJ. Effectiveness of progressive tendon-loading exercise therapy in patients with patellar tendinopathy: a randomised clinical trial. Br J Sports Med. 2021 May;55(9):501-509. doi: 10.1136/bjsports-2020-103403. Epub 2020 Nov 20. PMID 33219115
- [Background] Habets B, van Cingel REH, Backx FJG, van Elten HJ, Zuithoff P, Huisstede BMA. No Difference in Clinical Effects When Comparing Alfredson Eccentric and Silbernagel Combined Concentric-Eccentric Loading in Achilles Tendinopathy: A Randomized Controlled Trial. Orthop J Sports Med. 2021 Oct 27;9(10):23259671211031254. doi: 10.1177/23259671211031254. eCollection 2021 Oct. PMID 34722783
- [Background] Gravare Silbernagel K, Malliaras P, de Vos RJ, Hanlon S, Molenaar M, Alfredson H, van den Akker-Scheek I, Antflick J, van Ark M, Farnqvist K, Haleem Z, Kaux JF, Kirwan P, Kumar B, Lewis T, Mallows A, Masci L, Morrissey D, Murphy M, Newsham-West R, Norris R, O'Neill S, Peers K, Sancho I, Seymore K, Vallance P, van der Vlist A, Vicenzino B. ICON 2020-International Scientific Tendinopathy Symposium Consensus: A Systematic Review of Outcome Measures Reported in Clinical Trials of Achilles Tendinopathy. Sports Med. 2022 Mar;52(3):613-641. doi: 10.1007/s40279-021-01588-6. Epub 2021 Nov 19. PMID 34797533
- [Background] Habets B, van Cingel REH, Backx FJG, Huisstede BMA. Alfredson versus Silbernagel exercise therapy in chronic midportion Achilles tendinopathy: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Jul 11;18(1):296. doi: 10.1186/s12891-017-1656-4. PMID 28693535
- [Background] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396
- [Background] Schneebeli A, Falla D, Clijsen R, Barbero M. Myotonometry for the evaluation of Achilles tendon mechanical properties: a reliability and construct validity study. BMJ Open Sport Exerc Med. 2020 Feb 12;6(1):e000726. doi: 10.1136/bmjsem-2019-000726. eCollection 2020. PMID 32153987
- [Background] Nadeau MJ, Desrochers A, Lamontagne M, Lariviere C, Gagnon DH. Quantitative ultrasound imaging of Achilles tendon integrity in symptomatic and asymptomatic individuals: reliability and minimal detectable change. J Foot Ankle Res. 2016 Aug 17;9:30. doi: 10.1186/s13047-016-0164-3. eCollection 2016. PMID 27540416